CLINICAL TRIAL: NCT05399706
Title: Retrospective Cohort Analysis of Sex-specific Differences in Abdominal Aortic Aneurysm Complexity and Association With Adverse Outcomes
Brief Title: Sex-specific Differences in AAA Complexity
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Other Study IDs: 292985
Record Dates: First submitted 2022-05-24; First posted 2022-06-01 (Actual); Last update posted 2022-06-23 (Actual); Status verified 2022-06

CONDITIONS: AAA - Abdominal Aortic Aneurysm
MeSH Terms: conditions — Aortic Aneurysm, Abdominal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Men: Male participants
  Interventions: Diagnostic Test: CTA Aorta
- Women: Female Participants
  Interventions: Diagnostic Test: CTA Aorta

INTERVENTIONS:
Diagnostic Test: CTA Aorta — Computed Tomography Angiography - Aorta Whole

SUMMARY:
A retrospective cohort study of computed tomography scans of AAA patients considered for repair, in order to identify sex specific differences in abdominal aortic aneurysm (AAA) metrics and the association between anatomical differences/features of complexity and adverse patient outcome.

DETAILED DESCRIPTION:
A retrospective cohort study of computed tomography scans of AAA patients considered for repair.

The study aims to, firstly, identify sex specific differences in abdominal aortic aneurysm (AAA) metrics utilising manual and automated image processing techniques; and secondly, if numbers are sufficient, explore the association between features of AAA complexity and adverse patient outcome.

ELIGIBILITY:
Inclusion Criteria:

* All adult patients with AAA receiving assessment +/- primary open or endovascular repair at participating centre from 1/1/2010 to 31/12/2020.
* Must have AAA >= 5cm.
* Must have CT imaging within 1 year of operation or definitive turn down for treatment.

Exclusion Criteria:

* Insufficient CT imaging quality (>3mm slices) or lack of CT within 1 year of operation.
* Insufficient clinical data to establish risk factors or clinical outcomes.
* Ruptured aneurysm, aorto-iliac occlusive disease, isolated iliac aneurysm, penetrating aortic ulcer, dissection, juxta or supra-renal aneurysm.
* Secondary repair/not primary treatment decision for AAA repair.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with AAA receiving assessment +/- primary open or endovascular repair.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2022-07-31 (Estimated); Primary Completion 2024-10-01 (Estimated); Study Completion 2024-10-01 (Estimated)

PRIMARY OUTCOMES:
Sex-specific differences in thrombus burden | Pre-operative CT
  Volumetric assessment of aortic thrombus
Sex-specific differences in anatomical complexity | Pre-operative CT
  Anatomical as assessed by current IFU (instructions for use) criteria. (Anatomy within pre-specified vessel diameter, length, tortuosity and calcification criteria for insertion of endovascular stent graft for AAA repair.)

SECONDARY OUTCOMES:
Association between anatomical differences and adverse patient outcome for patients receiving operative repair - need for transfusion, risk of vessel injury, ischaemia (bowel or limb), renal injury and re-intervention/endoleak. | 30 days
  Post-operative outcomes

CONTACTS AND LOCATIONS:
Locations (1):
- Imperial College London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No